CLINICAL TRIAL: NCT05246566
Title: Assessment of Adults Epidemiological Characteristics of Status Epilepticus in the French West Indies and in French Guiana
Acronym: EpiDFA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Other Study IDs: 21_RIPH3-05
Record Dates: First submitted 2022-02-09; First posted 2022-02-18 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2023-10

CONDITIONS: Status Epilepticus; Epilepsy
Keywords: Status Epilepticus; Epilepsy; Epidemiology; Pronostic
MeSH Terms: conditions — Status Epilepticus; Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects covered for suspected or SE diagnosis: Patients covered for suspected or SE diagnosis defined by one of the following:
  * a prolonged generalized tonic-clonic crisis lasting more than 5 minutes and accompanied by impaired consciousness or at least 2 generalized tonic-clonic crisis without return to normal consciousness between crisis.
  * a focal convulsive crisis (motor or not) with disturbances of consciousness which lasts beyond 10 minutes or crisis which are repeated (≥ 2) at short intervals without recovery of interictal consciousness.
  * a focal convulsive crisis (motor or not) without alteration of consciousness that lasts beyond 10 to 15 minutes.
  * an absence-type crisis that lasts longer than 10 to 15 minutes.
  * a myoclonic, clonic and tonic crisis that lasts longer than 10 to 15 minutes.
  * a coma with an epileptic cause diagnosed on an EEG.
  Interventions: Other: Routine care

INTERVENTIONS:
Other: Routine care — The investigator takes care of the patient according to the protocol in force in his department and decides on the final orientation of the patient (transfer to intensive care unit/ICU, hospitalization or home discharge).
  No recommendations or instructions are given to the investigators. Each investigator is free to decide on his care and the terms of transfer, hospitalization and discharge.

SUMMARY:
The justification of this prospective and multicenter study is based on the absence of published data concerning, status epilepticus (SE), a pathology which seems frequent in the French West Indies (FWI) and French Guiana, and whose etiological and prognostic characteristics are often mentioned or assumed but which remain to be demonstrated. The scientific interest lies both in the knowledge of the epidemiology of this pathology and in the identification of the main etiologies, in particular the underlying brain lesions.

The morbidity of SE is significant, associating neurological disorders with impaired consciousness, respiratory, hemodynamic and cardiac rhythm disorders, as well as metabolic disorders such as acidosis. SE-related mortality in the acute phase ranges from 3-40% across studies and regions, while long-term mortality ranges from 17-80% depending on age, cause of SE, comorbidities and the occurrence of complications.

The prognosis of this pathology has however improved in recent years in developed countries or countries with a high level of health system. On the other hand, the morbidity and mortality of SE in the French overseas departments is not known, even if these territories are supposed to be at an equivalent level in terms of health system to that of mainland France.

DETAILED DESCRIPTION:
Epilepsy is a chronic neurological disease characterized by the occurrence of intermittent seizures, often isolated, but which can progress to status epilepticus (SE) when the seizures are repeated at short intervals without recovery of consciousness. SE is an acute complication that occurs during epileptic disease, but it can also occur outside of known epilepsy, indicative of acute neurological or systemic damage. SE is a neurological emergency, the second after stroke. The incidence of the occurrence of SE is estimated at 12.6 cases per 100,000 person-year, but is widely variable depending on the study region.

The epidemiological, clinical, etiological and prognostic characteristics of epilepsy and SE vary depending on the continent and region, mainly linked to the exposing or favoring factors as well as the socio-economic level of the population, the healthcare offer of the patient health system and accessibility to care for the population.

In France, the management of SE has been codified by Formalized Expert Recommendations (RFE) from learned societies in Emergencies and Resuscitation. The last updated RFE was published in 2018. However, very few studies have been carried out on SE in prehospital or emergencies department. There are no national epidemiological data on SE. To our knowledge, there is no data on the prevalence of SE in the French West Indies (FWI) and French Guiana and even less on the main aetiologies and prognosis of this acute neurological complication.

The interest of this prospective study is to evaluate, through the emergency system, the incidence, the modes of clinical presentation, the etiologies, the therapeutic modalities and finally the prognosis of SE in French overseas departments. This study is of scientific interest for the new knowledge it will bring, because there is no data concerning this relatively common pathology in these regions.

The results of the study would contribute to the improvement of scientific knowledge, to the highlighting of potential particularities and specificities of this pathology in the FWI and French Guiana, and would contribute to improving medical practice and the management of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years old) treated for SE by SAMU/SMUR and by emergencies or intensive care in the French West Indies and French Guiana.
* Covered for suspected or SE diagnosis defined by one of the following:

  * a prolonged generalized tonic-clonic crisis lasting more than 5 minutes and accompanied by impaired consciousness or at least 2 generalized tonic-clonic crisis without return to normal consciousness between crisis.
  * a focal convulsive crisis (motor or not) with disturbances of consciousness which lasts beyond 10 minutes or crisis which are repeated (≥ 2) at short intervals without recovery of interictal consciousness.
  * a focal convulsive crisis (motor or not) without alteration of consciousness that lasts beyond 10 to 15 minutes.
  * an absence-type crisis that lasts longer than 10 to 15 minutes.
  * a myoclonic, clonic and tonic crisis that lasts longer than 10 to 15 minutes.
  * a coma with an epileptic cause diagnosed on an EEG.
* Patient if he is able to, or representative of the patient in case of incapacity, having given his agreement for the use of his medical data for this research.

Exclusion Criteria:

* Age < 18 years old
* Absence of consent from the patient, or representative to the use of the data for the research.
* Patient whose main residence is not in the department where the study is taking place (vacationer for example).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients covered for suspected or SE diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 241 (Estimated)
Dates: Start 2022-05-15 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
To measure the annual incidence rate of occurrence of status epilepticus (SE) in adults treated by SAMU/SMUR and emergency services in the French West Indies and French Guiana. | 15 months
  The incidence rate of the occurrence of SE expressed per 100,000 person-years.This incidence rate will be calculated by dividing the number of new cases of SE during the 12 months of the inclusion phase of the study by the estimate of the average number of inhabitants aged 18 and over in each region of inclusion.

SECONDARY OUTCOMES:
To describe the epidemiological characteristics of status epilepticus in adults in the French West Indies and French Guiana in terms of patient profiles, associated factors, recurrences, causes and complications. | 15 months
  Characteristics of the patients (age, sex) / Number and percentage of patients with factors associated with SE (alcoholism, drug addiction, precarity, etc.) / Number and percentage of recurrences of SE episodes (antecedent of SE) / Number and percentage of the different causes causing a SE episode / Number and percentage of the different complications during the occurrence of a SE episode.

OTHER OUTCOMES:
To describe the neurological evolution 30 days and 90 days after the SE eoisode in adults in the French West Indies and French Guiana. | 15 months
  Number and percentage of patients with an unfavorable neurological evolution according to an assessment using the Modified Rankin Scale (MRS greater than 2) in the adult SE population at day 30 and day 90.
To measure the mortality rate at day 1, day 30 and day 90 after the onset of SE in adults treated by SAMU/SMUR and emergency services in the French West Indies and French Guiana. | 15 months
  Mortality rate in the adult SE population included in the study on day 1, day 30 and day 90.

CONTACTS AND LOCATIONS:
Overall Officials: Florian Negrello, MD, Principal Investigator — University Hospital Center of Martinique
Locations (4):
- France (4):
  - Hospital of Cayenne, Cayenne, French Guiana
  - Hospital of Basse-Terre, Basse-Terre, Guadeloupe
  - University Hospital Center of Guadeloupe, Pointe à Pitre, Guadeloupe
  - University Hospital Center of Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No